CLINICAL TRIAL: NCT03430661
Title: Single-center, Double-blind (ACT-246475), Open-label (Clopidogrel, Prasugrel, and Ticagrelor), Placebo-controlled, Randomized, Two-way Crossover Study to Investigate the Pharmacodynamics, Safety, and Tolerability of a Single Oral Dose of Clopidogrel or, Prasugrel, or Ticagrelor When Administered After a Single Subcutaneous Dose of the P2Y12 Antagonist ACT-246475 in Healthy Male and Female Subjects
Brief Title: A Study to Investigate the Interaction Between ACT-246475 and Clopidogrel, Prasugrel, and Ticagrelor in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ID-076-103
Record Dates: First submitted 2018-01-30; First posted 2018-02-13 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2022-11

CONDITIONS: Healthy
MeSH Terms: interventions — selatogrel; Clopidogrel; Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part A: Group 1 (Experimental): Clopidogrel will be administered 0.5 h after ACT-246475 or placebo, i.e., at the time of tmax
  Interventions: Drug: ACT-246475; Drug: Clopidogrel; Drug: Placebo
- Part A: Group 2 (Experimental): Clopidogrel will be administered 12 h after ACT-246475 or placebo
  Interventions: Drug: ACT-246475; Drug: Clopidogrel; Drug: Placebo
- Part A: Group 3 (Experimental): Any time interval up to 24 h between the administration of ACT-246475 or placebo and clopidogrel may be studied
  Interventions: Drug: ACT-246475; Drug: Clopidogrel; Drug: Placebo
- Part B: Group 1 (Experimental): Prasugrel will be administered 12 h after ACT-246475 or placebo
  Interventions: Drug: ACT-246475; Drug: Prasugrel; Drug: Placebo
- Part B: Group 2 (Experimental): Any time interval up to 24 h between the administration of ACT-246475 or placebo and prasugrel may be studied
  Interventions: Drug: ACT-246475; Drug: Prasugrel; Drug: Placebo
- Part B: Group 3 (Experimental): Any time interval up to 24 h between the administration of ACT-246475 or placebo and prasugrel may be studied
  Interventions: Drug: ACT-246475; Drug: Prasugrel; Drug: Placebo
- Part C: Group 1 (Experimental): Ticagrelor will be administered 0.5 h after ACT-246475 or placebo, i.e., at the time of tmax
  Interventions: Drug: ACT-246475; Drug: Placebo; Drug: Ticagrelor
- Part C: Group 2 (Experimental): Any time interval up to 24 h between the administration of ACT-246475 or placebo and ticagrelor may be studied
  Interventions: Drug: ACT-246475; Drug: Placebo; Drug: Ticagrelor
- Part C: Group 3 (Experimental): Any time interval up to 24 h between the administration of ACT-246475 or placebo and ticagrelor may be studied
  Interventions: Drug: ACT-246475; Drug: Placebo; Drug: Ticagrelor

INTERVENTIONS:
Drug: ACT-246475 — Lyophilized ACT-246475A to be reconstituted with 1 mL of water for injection
Drug: Clopidogrel — Tablet for oral administration (300 or 600 mg)
  Arms: Part A: Group 1; Part A: Group 2; Part A: Group 3
Drug: Prasugrel — Tablet for oral administration (60 mg)
  Arms: Part B: Group 1; Part B: Group 2; Part B: Group 3
Drug: Placebo — Matching ACT-246475 placebo will consist of sterile 0.9% w/v sodium chloride solution
Drug: Ticagrelor — Tablet for oral administration (180 mg)
  Arms: Part C: Group 1; Part C: Group 2; Part C: Group 3

SUMMARY:
The primary objective of this study is to assess the pharmacodynamic (PD) effects of clopidogrel, prasugrel, and ticagrelor when administered after a single subcutaneous (s.c.) dose of ACT-246475 in healthy male and female subjects

ELIGIBILITY:
Main Inclusion Criteria:

* Signed informed consent
* Healthy male and female subjects aged between 18 and 65 years (inclusive) at screening
* Body mass index of 18.0 to 31.0 kg/m2 (inclusive) at Screening
* Women of childbearing potential must have a negative serum pregnancy test and use reliable birth controls from screening up to at least 30 days after last study treatment administration
* Systolic blood pressure (SBP) 100-140 mmHg, diastolic blood pressure (DBP) 50-90 mmHg, and pulse rate 50-90 beats per minute (bpm) (inclusive) at screening
* Healthy on the basis of physical examination, cardiovascular assessments, and laboratory tests
* Maximum (at peak) platelet aggregation ≥ 40% (light transmission aggregometry [LTA]) upon 20 μM adenosine diphosphate (ADP) activation at screening
* Values of closure time tested with the Platelet Function Analyzer (PFA) equipment, for both cartridges of collagen/adrenaline and collagen/ADP below the upper limit of normal range at screening

Main Exclusion Criteria:

* Pregnant or lactating women
* Known hypersensitivity to ACT-246475, clopidogrel, prasugrel, ticagrelor, any of their excipients, or drugs of the same class
* Any contraindication to clopidogrel, prasugrel, or ticagrelor treatment
* Known hypersensitivity or allergy to natural rubber latex
* Platelet count < 120 × 109 L-1 at Screening and Day -1
* Known platelet disorders (e.g., Glanzmann thromboasthenia, von Willebrand disease, platelet release defect)
* Previous treatment with acetylsalicylate, non-steroidal anti-inflammatory drugs, P2Y12 receptor antagonists, or any medication with blood-thinning activity (i.e., injectable or oral anticoagulants) within 3 weeks prior to study treatment administration
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Time-matched comparisons of IPA% (MPA) between treatments (i.e., Treatment A1 vs A2, Treatment B1 vs B2, and treatment C1 vs C2, treatments are defined below) following administration of ACT-246475 and its matching placebo. | From baseline up to 48 hours
  - IPA%[MPA] will be calculated as mean change in percentage from baseline for each time point.
Time-matched comparisons of IPA %(PRU) between treatments (i.e., Treatment A1 vs A2, Treatment B1 vs B2, and treatment C1 vs C2) following administration of ACT-246475 and its matching placebo. | From baseline up to 48 hours
  - IPA%[PRU] will be calculated as mean change in percentage from baseline for each time point.
  Treatment A1: single s.c. dose administration of ACT-246475-matching placebo followed by a single oral dose of clopidogrel (600 mg).
  Treatment A2: single s.c. dose administration (16 mg) of ACT-246475 followed by a single oral dose of clopidogrel (300 mg).
  Treatment B1: single s.c. dose administration of ACT-246475-matching placebo followed by a single oral dose of prasugrel (60 mg).
  Treatment B2: single s.c. dose administration (16 mg) of ACT-246475 followed by a single oral dose of prasugrel (60 mg).
  Treatment C1: single s.c. dose administration of ACT-246475-matching placebo followed by a single oral dose of ticagrelor (180 mg).
  Treatment B2: single s.c. dose administration (16 mg) of ACT-246475 followed by a single oral dose of ticagrelor (180 mg).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (1):
- Biotrial Inc, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schilling U, Dingemanse J, Dobrow M, Baumann M, Riederer MA, Juif PE, Ufer M. Insights from In Vitro and Clinical Data to Guide Transition from the Novel P2Y12 Antagonist Selatogrel to Clopidogrel, Prasugrel, and Ticagrelor. Thromb Haemost. 2021 Jun;121(6):755-766. doi: 10.1055/s-0040-1721773. Epub 2021 Jan 7. PMID 33412611